CLINICAL TRIAL: NCT05016271
Title: Health Benefits of Air Purifiers in Primary School Students: A Randomized Controlled Trial
Brief Title: Health Benefits of Air Purifiers in Primary School Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FDUEH-7
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cardiopulmonary Function; Child
Keywords: Air pollution; Particulate matter; Air Purifiers; Cardiopulmonary system
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True air purifier group (Experimental): Children in this group will receive an intervention of air purifiers with high-efficiency particulate air (HEPA) filters.
  Interventions: Behavioral: Air purifier and fresh air ventilation systems with high-efficiency particulate air (HEPA) filters
- Sham air purifier group (Sham Comparator): Children in this group will receive an intervention of air purifiers without high-efficiency particulate air (HEPA) filters.
  Interventions: Behavioral: Air purifier and fresh air ventilation systems without high-efficiency particulate air (HEPA) filters

INTERVENTIONS:
Behavioral: Air purifier and fresh air ventilation systems with high-efficiency particulate air (HEPA) filters — This group will receive an intervention of true air purifiers. The air purifiers in classroom (air purifiers and fresh air ventilation systems with HEPA filters) will operate during the school time and the air purifiers in bedrooms (air purifiers with HEPA filters) operate during the home time in the intervention period (4 months anticipated).
  Arms: True air purifier group
Behavioral: Air purifier and fresh air ventilation systems without high-efficiency particulate air (HEPA) filters — This group will receive an intervention of sham air purifiers. The air purifiers in classroom (air purifiers and fresh air ventilation systems without HEPA filters) will operate during the school time and the air purifiers in bedrooms (air purifiers without HEPA filters) operate during the home time in the intervention period (4 months anticipated).
  Arms: Sham air purifier group

SUMMARY:
This study aims to explore changes in cardiopulmonary function and other health indicators in primary school students with the intervention of air purifiers on a randomized controlled trial.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial among 110 healthy children in Jiaozuo city, Henan, China. The eligible children will be divided into two groups according to their classes and randomly receive interventions of either true or sham air purifiers. The air purifiers devices in classroom [air purifiers and fresh air ventilation systems] will operate during the school time and the devices in bedrooms (air purifiers) operate during the home time in the intervention period. All the participants and investigators will be blinded to the group assignment. Epidemiological questionnaires (i.e., basic characteristics, eating habits, daily schedule, etc.) will be conducted and health indicators (i.e., blood pressure, pulmonary function indicators, fractional exhaled nitric oxide, and fractional exhaled carbon monoxide) and biological specimens (i.e., morning urine, venous blood, exhaled breath condensate, and feces) will be evaluated and collected at baseline and after the completion of intervention period (4 months anticipated).

ELIGIBILITY:
Inclusion Criteria:

* Age of between 8 and 12 years old
* Males and female of ethnic Han
* Subjects who have no plans to change classroom during the intervention period
* Subjects who staying in Jiaozuo city during the intervention period

Exclusion Criteria:

* Subjects with asthma, childhood diabetes, childhood hypertension, and behavioral disorders
* Subjects who plan to transfer or move offsite within six months
* Subjects who decorated or plan to decorate home within six months
* Subjects with smokers in the household

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of heart rate variability | Baseline and after the completion of intervention period (4 months anticipated)
  Nihon Kohden Electrocardiograph and Carepatch Electrocardiogram are used to measure heart rate variability, including standard deviation of all normal-to-normal R-R intervals (SDNN), standard deviation of sequential five-minute R-R interval means (SDANN), root-mean-square difference of successive normal R-R intervals (RMSSD), low frequency (LF), and high frequency (HF) in intervention and control groups. To eliminate possible errors, measurements are conducted by the same trained staff using the same instrument.
Changes of forced expiratory volume in 1 s (FEV1) | Baseline and after the completion of intervention period (4 months anticipated)
  The pulmonary function measures are performed by the professional medical device. Before the pulmonary function test, subjects practice several times with the guidance of professional staff. During the examination, each subject in a sitting position and clamp the nose clip, and repeat the test, with the best result as the criterion.
Changes of forced vital capacity (FVC) | Baseline and after the completion of intervention period (4 months anticipated)
  The pulmonary function measures are performed by the professional medical device. Before the pulmonary function test, subjects practice several times with the guidance of professional staff. During the examination, each subject in a sitting position and clamp the nose clip, and repeat the test, with the best result as the criterion.
Changes of forced expiratory volume in 1 s (FEV1) / forced vital capacity (FVC) ratio | Baseline and after the completion of intervention period (4 months anticipated)
  The pulmonary function measures are performed by the professional medical device. Before the pulmonary function test, subjects practice several times with the guidance of professional staff. During the examination, each subject in a sitting position and clamp the nose clip, and repeat the test, with the best result as the criterion.
Changes of peak expiratory flow (PEF) | Baseline and after the completion of intervention period (4 months anticipated)
  The pulmonary function measures are performed by the professional medical device. Before the pulmonary function test, subjects practice several times with the guidance of professional staff. During the examination, each subject in a sitting position and clamp the nose clip, and repeat the test, with the best result as the criterion.
Changes of fractional exhaled nitric oxide (FeNO) levels | Baseline and after the completion of intervention period (4 months anticipated)
  A NIOX VERO Sensor is used to measure fractional exhaled nitric oxide (FeNO) as a biomarker for airway inflammation. After deep breathing, the subjects gently inhaled into the device. The instrument shows FeNO level of the subjects.
Changes of fractional exhaled carbon monoxide (FeCO) levels | Baseline and after the completion of intervention period (4 months anticipated)
  Use PICO to measure fractional exhaled carbon monoxide (FeCO) as a biomarker for cardiovascular risk. After deep breathing and holding the breath for 15 seconds, the subjects gently inhaled into the device. The instrument shows FeCO level of the subjects.
Changes of blood pressure | Baseline and after the completion of intervention period (4 months anticipated)
  Using Omron blood pressure monitor to measure the systolic blood pressure (SBP), diastolic blood pressure (DBP), and pulse pressure for each subject by the trained staff using the same instrument.

SECONDARY OUTCOMES:
Changes of C-reactive protein (CRP) | Baseline and after the completion of intervention period (4 months anticipated)
  Detect the concentration of C-reactive protein (CRP) in blood sample to examine the different level of inflammation between the groups of intervention and control.
Changes of 8-hydroxydeoxyguanosine (8-OHdG) | Baseline and after the completion of intervention period (4 months anticipated)
  Detect the concentration of 8-hydroxydeoxyguanosine (8-OHdG) in urine sample of groups of intervention and control. 8-OHdG is a biomarker for DNA oxidative damage.
Changes of persistent response (PR) | Baseline and after the completion of intervention period (4 months anticipated)
  Examine persistent response (PR) as the index to test the focus ability of children. The test is performed by the Wisconsin Card Sorting Test (WCST) through a computer, and the index reflects the ability of cognitive transfer. The normal value is less than or equal to 27.
Differences in metabolite levels detected in metabolomics between groups of intervention and control. | Baseline and after the completion of intervention period (4 months anticipated)
  Mass spectrometry-based serum metabolomics is non-targeted. The study is to explore the differential metabolites in blood/urine/exhaled breath condensate (EBC) samples of the groups of intervention and control.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided